CLINICAL TRIAL: NCT00657540
Title: A Phase III Multicenter Clinical Trial of Analatro® [Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2] in Patients With Systemic Latrodectism
Brief Title: Black Widow Spider Antivenin for Patients With Systemic Latrodectism
Acronym: BWSP3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: Rare Disease Therapeutics Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XF-07/03
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Latrodectism
Keywords: black widow spider; antivenom; latrodectism
MeSH Terms: conditions — Spider Bites | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Analatro (Experimental): Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2
  Interventions: Drug: Analatro
- Normal Saline Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Analatro — 30 mL of lyophilized antivenom, reconstituted in 50 mL saline infused over 10 minutes, up to 2 doses
  Arms: Analatro
Drug: Saline — 50 mL of saline infused over 10 minutes
  Other Names: Placebo
  Arms: Normal Saline Placebo

SUMMARY:
The purpose of this study is to test the efficacy and safety of a new antivenom called Analatro® for treating black widow spider bites in patients who present to a hospital emergency room within 24 hours of symptom onset. This study will be a phase III, multi-center, double-blind, randomized controlled study that takes place in emergency departments. The primary aim of this study is to determine the proportion of patients in which pain control was not achieved by 48 hours post treatment. Secondary aims are as follows: 1) a reduction in pain intensity at the end of the treatment phase compared to baseline; 2) the proportion of patients with a clinically significant decrease in pain intensity at 30 minutes post-treatment; 3) the proportion of patients in which drug-related adverse events occurred; and 4) to determine if serious, drug-related adverse events in Analatro-treated patients occurred at a rate greater than one in 10 (10%).

DETAILED DESCRIPTION:
Instituto Bioclon S.A. de C.V. has developed Analatro®, an antibody fragment (Fab2) containing widow spider (Latrodectus) antivenom, and proposes to conduct a clinical trial in hospital emergency departments to assess the efficacy and safety of this product in patients with moderate to severe pain associated with Latrodectus envenomation (latrodectism). The primary objectives of this Phase III, multi-center, double-blind, controlled study are as follows:

To determine the efficacy of Analatro compared to control for the treatment of latrodectism as measured by the proportion of patients in whom pain control is not achieved (e.g., treatment failure)

To further characterize the safety profile of Analatro, including comparison of the rate of drug-related adverse events to control for the treatment of latrodectism

The flow of study procedures are illustrated in the chart on the following page. All patients who consent to participate will be given a visual analog scale (VAS, 0=no pain to 100mm=worst possible pain) for assessing pain intensity. Patients that meet all study enrollment requirements, including a minimum age of 10 years, a clinical diagnosis of latrodectism and a VAS pain score of ≥40 mm (moderate to severe pain) will be randomly assigned to be treated with Analatro or control. A screening phase will be completed, during which time preliminary procedures will be performed by the investigator (medical history, physical exam, and pregnancy test as applicable) and two doses of Analatro or two doses of saline control will be prepared. Fentanyl may be administered intravenously as needed for pain relief during the screening phase at a dosage not to exceed 1.5 µg/kg/hr. At the end of the screening phase, baseline measurements (vital signs, VAS pain score) will be performed. Patients must have a baseline VAS score ≥40 mm to receive study medication.

Eligible patients will begin a 2.5 hour treatment phase. Dose 1 of study medication (50 mL) will be infused intravenously over 10 minutes. Thirty minutes after the start of Dose 1, pain intensity will be assessed (VAS2), vital signs will be recorded (VS2), and a blood sample collected (B2). Clinical improvement in this study will be defined as a VAS score that is at least 13mm less than the baseline VAS score (VAS1). Patients that fail to show clinical improvement at 30 minutes will receive Dose 2 of study medication (Dose 2 will be identical to Dose 1). Patients showing clinical improvement will not receive Dose 2.

Thirty minutes after VAS2 (or after the start of Dose 2, if applicable), VAS3 will be administered, vital signs (VS3) will be recorded, and a blood sample (B3) will be collected. If the patient has not clinically improved relative to baseline, the patient will be deemed a treatment failure; the treatment phase will be discontinued, and the patient will be treated in accordance with standard of care by the investigator and/or treating physician. Patients that have clinically improved will remain in the treatment arm.

The remaining 1.5 hours of the treatment arm will consist of serial assessments of pain intensity (VAS4, 5 and 6), vital signs (VS4, 5 and 6), and collection of one blood sample (B4, 5 and 6) every 30 minutes. After each VAS, the patient must continue to show clinical improvement relative to baseline to remain in the treatment arm. Otherwise, the patient will exit the treatment phase and be treated in accordance with standard of care. No analgesics will be allowed during the treatment phase to eliminate the potential confounding effect of pain medication on assessing the effectiveness of the study medication on clinical improvement. Routine decision points for treatment failure (every thirty minutes) will promote accurate identification of treatment failures without compromising timely provision of pain medication in absence of clinical improvement.

All patients will be closely monitored for adverse events during Dose 1 of treatment until the time of discharge from the emergency department. Follow-up for possible adverse events and recurring/residual symptoms will be conducted by telephone on Days 2, 10, and 17 after discharge from the emergency department.

Treatment failure will be defined as (1) early exit from the treatment phase due to absence of clinical improvement relative to baseline and/or (2) patient requires prescription pain medication or Antivenin Latrodectus Mactans (Merck) for pain associated with the study condition being treated at any time after the treatment phase up to 48 hours after the time of discharge from the emergency department. To improve accurate identification of treatment failure after discharge, no preventative pain medication will be administered or prescribed to patients that successfully complete the treatment phase. Patients will be encouraged to call the investigator or return to the emergency department, if necessary, for proper evaluation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain intensity measured using the visual analog scale (VAS score ≥ 40mm) at the start of screening phase (VAS 0)
* Diagnosis of latrodectism by the Investigator, with concurrence of diagnosis by a physician not directly involved with the study
* Moderate to severe pain intensity measured using the visual analog scale (VAS score ≥ 40mm) at Baseline (VAS 1)

Exclusion Criteria:

* Less than 10 years of age
* Presents to the emergency department of any healthcare facility greater than 24 hours after onset of symptoms
* Has a known (self-reported) hypersensitivity to fentanyl, morphine, diazepam, or equine serum
* History of significant cardiac, respiratory, hepatic or renal disease, psychiatric disorder or chronic pain syndrome that in the investigator's assessment would confound efficacy or safety endpoint assessment (e.g., a bite to the leg of a patient with reflex sympathetic dystrophy)
* History or suspected history or substance abuse
* Pregnant or breast-feeding
* Has a distracting injury with acute pain, or is unable to make a reliable self-report of pain intensity to pain relief based solely on the condition of interest
* Was already treated with Merck Antivenin Latrodectus Mactans for signs/symptoms related to the current widow spider bite
* Unable to provide a telephone number to be contacted for follow-up interviews on Days 2, 10, and 17 after discharge from the emergency department

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Dart, MD, PhD, Principal Investigator — Rocky Mountain Poison & Drug Center - Denver Health; Walter Garcia, MD, Study Director — Instituto Bioclon S.A. de C.V.
Locations (16):
- United States (16):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Maricopa Medical Center, Phoenix, Arizona
  - University of California Davis, Davis, California
  - University California San Francisco - Fresno, Fresno, California
  - University of California Irvine, Irvine, California
  - Loma Linda University, Loma Linda, California
  - University of California San Diego, San Diego, California
  - San Diego Children's Hospital, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Cape Coral Hospital, Cape Coral, Florida
  - University of Florida, Department of Emergency Medicine, Gainesville, Florida
  - LSU Health Sciences, Shreveport, Louisiana
  - University of New Mexico, Albuquerque, New Mexico
  - Texas Tech - West Texas Regional Poison Center, El Paso, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dart RC, Bush SP, Heard K, Arnold TC, Sutter M, Campagne D, Holstege CP, Seifert SA, Lo JCY, Quan D, Borron S, Meurer DA, Burnham RI, McNally J, Garcia-Ubbelohde W, Anderson VE. The Efficacy of Antivenin Latrodectus (Black Widow) Equine Immune F(ab')2 Versus Placebo in the Treatment of Latrodectism: A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial. Ann Emerg Med. 2019 Sep;74(3):439-449. doi: 10.1016/j.annemergmed.2019.02.007. Epub 2019 Mar 27. PMID 30926190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the nature of the treatment emergent condition of interest, no patients were actively recruited. Potential subjects presenting with moderate to severe pain associated with diagnosed latrodectism were evaluated at 16 sites across the United States. The first subject was enrolled on 10/08/09. The last subject completed the study on 10/27/14.
Groups:
- Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2: Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2
  Analatro: 30 mL of lyophilized antivenom, reconstituted in 50 mL saline infused over 10 minutes, up to 2 doses
- Normal Saline: Normal Saline
  Saline: 50 mL of saline infused over 10 minutes
Period: Overall Study
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline
Started | 29 | 31
Completed | 28 (All subjects had a known treatment failure disposition at time of loss to follow-up.) | 27 (All subjects had a known treatment failure disposition at time of loss to follow-up.)
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Population: The analysis population consists of all patients that were randomized and received any study drug (modified intent-to-treat population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (15.18) | 41.0 (17.84) | 39.2 (16.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 18 | 23 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 17 | 30
  Not Hispanic or Latino | 16 | 14 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 20 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 11 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 31 | 60
Baseline VAS Pain Score (mm) [Mean (Standard Deviation); unit: mm] — The Visual Analog Scale (VAS) ranged from 0 (no pain) to 100 mm (worst possible pain).
  mm | 79.7 (13.16) | 73.8 (16.14) | 76.7 (14.96)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure
Description: The primary efficacy endpoint for this study was the number of subjects in which pain control was not achieved 48 hours post-study drug infusion as identified by treatment failure. A treatment failure was defined as a subject who did not achieve pain control during the treatment phase, up to 48 hours after Dose 1 infusion start time. Subjects were deemed treatment failures if they met one or more of the following criteria:
  * Subject did not complete the treatment phase due to absence of clinically significant improvement in pain intensity relative to baseline at 60, 90, 120, or 150 minutes post start of Dose 1.
  * Subject required treatment with commercially available antivenin or prescription pain medication for signs and symptoms associated with latrodectism at any time during the treatment phase up to 48 hours after Dose 1 infusion start time.
Time Frame: From start of Dose 1 infusion to 48 hours post treatment
Population: The analysis population consists of all subjects that were randomized and received any study drug (modified intent to treat population).
Measure: Count of Participants; unit: Participants
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline
Number analyzed (Participants) | 29 | 31
Participants | 15 | 24
Statistical Analysis 1: Comparison: Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 vs Normal Saline; Test type: Superiority or Other; p = 0.0185, Chi-squared; The proportion of treatment failures was compared between groups using a one-sided test at the 0.025 level of significance

2. Secondary Outcome: Number of Participants With at Least 13 mm Reduction in Pain Score at 30 Minutes Post-Treatment
Description: The number of patients with a clinically significant decrease in pain intensity at 30 minutes post-treatment (after Dose 1 and Dose 2, as applicable) will be measured by the patient's self-assessment of pain intensity using the visual analog scale (VAS). A clinically significant reduction in pain is defined as a decrease in VAS scores of greater than or equal to 13 mm. The VAS ranged from 0 (no pain) to 100 mm (worst possible pain).
Time Frame: 30 minutes post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline
Number analyzed (Participants) | 29 | 31
Participants | 13 | 11
Statistical Analysis 1: Comparison: Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 vs Normal Saline; Test type: Superiority or Other; p = 0.2302, Chi-squared; Chi-squared tests at the 0.025 level of significance were used to test for a difference in proportions between the treatment groups

3. Secondary Outcome: Drug-related Adverse Events
Description: To evaluate safety of Analatro, the number of subjects experiencing at least one adverse event (AE) that was determined to be related to study drug was computed for each treatment group. All AEs classified as definitely or possibly related to study drug were considered drug-related.
Time Frame: Start of Dose 1 through 17 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline
Number analyzed (Participants) | 29 | 31
Participants | 16 | 18
Statistical Analysis 1: Comparison: Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 vs Normal Saline; Test type: Superiority or Other; p = 0.8213, Chi-squared; The proportion of subjects with at least one drug-related adverse event by treatment groups using a two-sided test at the 0.05 level of significance

4. Secondary Outcome: Number of Participants With at Least 13 mm Reduction in Pain Score at Any Time Point
Description: The number of patients with a clinically significant decrease in pain intensity relative to baseline at any time point during the treatment phase was measured by the patient's self-assessment of pain intensity using the visual analog scale (VAS). A clinically significant reduction in pain was defined as a decrease in VAS scores of greater than or equal to 13 mm. The VAS ranged from 0 (no pain) to 100 mm (worst possible pain).
Time Frame: Start of Dose 1 to any post-infusion time point
Measure: Count of Participants; unit: Participants
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline
Number analyzed (Participants) | 29 | 31
Participants | 19 | 18
Statistical Analysis 1: Comparison: Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 vs Normal Saline; Test type: Superiority or Other; p = 0.2765, Chi-squared; The proportion of subjects with decreased pain at any time point between treatment groups using a one-sided test at the 0.025 level of significance

5. Secondary Outcome: Drug-related Serious Adverse Events
Description: The number of subjects with drug-related serious adverse events.
Time Frame: Start of Dose 1 through 17 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events from the time of consent through 17 days post start of Dose 1.
Arm/Group | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/31
Other Adverse Events (participants affected / at risk) | 26/29 | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 (N=29) | Normal Saline (N=31)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — A subject was hospitalized for the treatment of cellulitis after receiving placebo. The subject had a previous history of methicillin-resistant staphylococcus aureus related to cellulitis. The event was determined to be not related to study drug.
Inadequate Pain Control (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — A subject was hospitalized for inadequate pain control 24 hours after receiving placebo. The subject was treated with analgesics and was discharged after 3 days of hospitalization. This event was determined to not be related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2 (N=29) | Normal Saline (N=31)
Constipation (Gastrointestinal disorders) | 0 | 6
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Chills (General disorders) | 3 | 7
Fatigue (General disorders) | 1 | 2
Inflammation (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3
Headache (Nervous system disorders) | 5 | 4
Paraesthesia (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 17
Rash (Skin and subcutaneous tissue disorders) | 4 | 8
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study is limited by the small sample size; however this trial was powered appropriately for an orphan indication. The study is also limited by the difficulty in confirming latrodectism without a spider or clear history of seeing a spider.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No